CLINICAL TRIAL: NCT06402526
Title: Unicentre Parallel Open Randomized Trial to Evaluate the Efficacy of a Mobile Epilepsy Education Application Developed For The Parents/Caregivers of Children With Epilepsy in Canada
Brief Title: Evaluating the Efficacy of a Mobile Epilepsy Education Application
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Collaborators: The Scientific and Technological Research Council of Turkey (Other)
Responsible Party: Principal Investigator, Kenneth Myers, MD, Principal Investigator, McGill University Health Centre/Research Institute of the McGill University Health Centre
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: MEA-EE (2024-10228)
Record Dates: First submitted 2024-04-29; First posted 2024-05-07 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2024-06

CONDITIONS: Epilepsy; Epilepsy in Children; Anxiety; Knowledge, Attitudes, Practice
Keywords: Epilepsy; Mobile application; Education; Anxiety; Knowledge; Parents/Caregivers
MeSH Terms: conditions — Epilepsy; Anxiety Disorders; Behavior

STUDY DESIGN:
Intervention Model Description: Eligible participants will be randomly allocated in a 1:1 ratio to the intervention group (use of MEEP) or the control group (standard care).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Mobile Epilepsy Education Package (Experimental): The Mobile Epilepsy Education Package (MEEP) consists of 2 parts. The first part entails the delivery of the "MEEP education", and the second part consists of the "Parental Monitoring Section". The intervention group will use MEEP for 4 weeks.
  Interventions: Other: Mobile Epilepsy Education Package
- Standard care consisting of epilepsy education (Other): Standard care consisting of epilepsy education and support offered at the study setting by members of the Pediatric Neurology Clinic was chosen as the comparator and serves as the control group.
  Interventions: Other: Standard care consisting of epilepsy education

INTERVENTIONS:
Other: Mobile Epilepsy Education Package — MEEP education section contains a range of topics. After completing the relevant section at the end of each week, participants complete the end-of-section test and switch to the next week's topic. Completion of the first part will take approximately 90-120 minutes per week for a total of 4 weeks of use.
  Parental Monitoring Section, parents can actively record information on the mobile application related to their child's diagnosis (anonymous); treatments; timing and frequency of the seizures; and appointments; and schedule treatment and examination reminders to optimize compliance. Completion of this second part will take approximately 1-2 minutes and depends on the parental choice to use and how much information they would like to share. The second part, together with the first part, will be evaluated for a total of 1 month.
  Arms: Mobile Epilepsy Education Package
Other: Standard care consisting of epilepsy education — This standard care includes the information and education provided by nurses and physicians during visits and hospitalisations. Standard information and education include topics such as: counseling by the neurologist regarding seizure safety precautions, prognosis, and sudden unexpected death in epilepsy (SUDEP); provision of paper or electronic resources regarding epilepsy; and telephone support provided by neurology clinic nurse regarding any issues or concerns). Information and education is usually provided orally and through printed brochures.
  Arms: Standard care consisting of epilepsy education

SUMMARY:
Background. Following a childhood diagnosis of epilepsy, children and their families encounter significant concerns about the disease trajectory, side effects of anti-seizure medications, and long-term prognosis. The multitude of uncertainties can cause significant anxiety in the family, often within the context of limited supports and resources. Epilepsy education can help address these concerns, mitigating the development of anxiety, ultimately leading to better patient-, family- and system-level outcomes. Globally, the MEEP is the only mobile application providing education, monitoring of symptoms, and tracking of medical appointments. The original MEEP was developed, tested, and integrated into practice in Turkey; the investigators will now evaluate the efficacy of an English and French version of the MEEP for families of children with epilepsy in Canada.

A two-group, single-center, randomized controlled intervention trial with 1:1 allocation ratio will be conducted in the Pediatric Neurology Clinic of the Montreal Children's Hospital. Seventy-two caregivers of children with epilepsy (intervention=36, control= 36), aged 1-17 years and treated at the study site will be eligible. Family Introduction Form, Epilepsy Information Scale for Parents and Parental Anxiety Scale for Seizures will be used to collect data at baseline and 3 weeks post-delivery of the 7-week intervention. The MEEP consists of 2 parts. The first part entails the delivery of the educational content of the MEEP, and the second part consists of a "Parental Monitoring Section." Comparator. The control group will continue to benefit from the standard educational services provided by the study site.

DETAILED DESCRIPTION:
OBJECTIVES:

Evaluate the efficacy of an English and French version of the Mobile Epilepsy Education Package (MEEP) for parents/caregivers of children with epilepsy in Canada.

Primary Objective:

To determine whether the MEEP used by parents/caregivers with children diagnosed with epilepsy increases the level of knowledge about epilepsy.

Secondary Objectives

1. To determine whether MEEP used by parents/caregivers of children with epilepsy reduces their anxiety about epilepsy.
2. To determine whether there is an increase in adherence to treatment by using the following MEEP features:

   1. "treatment/exam control time reminder" tab in the "follow-up section" of MEEP; and
   2. data on app usage (number of logins, time spent on app).

Primary and Secondary Endpoints/Outcome Measures The primary outcome is epilepsy knowledge and will be assessed using the " Epilepsy Knowledge Scale for Parents." The secondary outcome is parental anxiety and will be assessed with the "Parental Anxiety Scale for Seizures."

Other secondary outcomes are:

1. To determine whether there is an increase in adherence to treatment by using the "treatment/exam control time reminder" tab in the "follow-up section" of MEEP.
2. To determine whether there is an increase in adherence to treatment by using the data on app usage (number of logins, time spent on app).

ELIGIBILITY:
Inclusion Criteria:

* Parents/caregivers whose children are between 1-17 years old;
* Parents/caregivers whose child was diagnosed with epilepsy at least 2 months ago;
* At least one primary caregiver is comfortable interacting in English or French; and
* At least one primary caregiver owns and uses a smartphone on a daily basis.

Exclusion Criteria:

- Inability to provide informed consent for any reason.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2024-06-10 (Actual); Primary Completion 2024-08-30 (Actual); Study Completion 2024-12-30 (Actual)

PRIMARY OUTCOMES:
Change in epilepsy knowledge after 1 month of use of the Mobile Epilepsy Education Package | 7 weeks
  This will be assessed using the "Epilepsy Knowledge Scale for Parents." This scale consists of 20 questions including the cause of seizures, emergency care, complications of seizures, cognitive and psychosocial consequences and limitations. In scoring the items in the scale, False means "0" and True means "1". A score between 0-20 can be obtained from the scale. A high total score indicates that parents have a high level of knowledge about epilepsy.

SECONDARY OUTCOMES:
Change in epilepsy anxiety after 1 month of use of the Mobile Epilepsy Education | 7 weeks
  This will be assessed with the "Parental Anxiety Scale for Seizures." This scale consists of 9 items in 5-point Likert type. Each item in the scale is scored between 1 and 5. A score between 9 and 45 can be obtained from the scale. A high total score indicates that parents have low anxiety about seizures.

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Alexis Myers, MD PhD FRCPC, Principal Investigator — RI-MUHC, Montreal Children's Hospital, McGill University; Dilek Sayik, RN, PhD, Study Chair — Ingram School of Nursing, McGill University; Ayfer Acikgoz, RN, PhD, Study Chair — Faculty of Health Sciences, Eskisehir Osmangazi University; Argerie Tsimicalis, RN, PhD, Study Chair — Shriners Hospitals for Children, Ingram School of Nursing, McGill University
Locations (2):
- Canada (2):
  - Montreal Children's Hospital, Montreal, Quebec
  - Research Institute of the McGill University Health Centre, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: Yes
Share study protocol, materials (eg consent form, recruitment flyers). App will be available in the future for free download.
Supporting Information: Study Protocol, SAP
Time Frame: It is completed December 2024.
Access Criteria: The study protocol will be published in a journal. ICF can be requested from the author.

REFERENCES:
- [Result] Aaberg KM, Gunnes N, Bakken IJ, Lund Soraas C, Berntsen A, Magnus P, Lossius MI, Stoltenberg C, Chin R, Suren P. Incidence and Prevalence of Childhood Epilepsy: A Nationwide Cohort Study. Pediatrics. 2017 May;139(5):e20163908. doi: 10.1542/peds.2016-3908. Epub 2017 Apr 5. PMID 28557750
- [Result] Austin J, Dunn D, Huster G, Rose D. Development of scales to measure psychosocial care needs of children with seizures and their parents. 1. J Neurosci Nurs. 1998 Jun;30(3):155-60. doi: 10.1097/01376517-199806000-00002. PMID 9689606
- [Result] Austin JK, McNelis AM, Shore CP, Dunn DW, Musick B. A feasibility study of a family seizure management program: 'Be Seizure Smart. Journal of Neuroscience Nursing. 2002; 34(1): 30.
- [Result] Bakula DM, Wetter SE, Peugh JL, Modi AC. A Longitudinal Assessment of Parenting Stress in Parents of Children with New-Onset Epilepsy. J Pediatr Psychol. 2021 Jan 20;46(1):91-99. doi: 10.1093/jpepsy/jsaa091. PMID 33053164
- [Result] Carlson JM, Miller PA. Family burden, child disability, and the adjustment of mothers caring for children with epilepsy: Role of social support and coping. Epilepsy Behav. 2017 Mar;68:168-173. doi: 10.1016/j.yebeh.2017.01.013. Epub 2017 Feb 12. PMID 28199920
- [Result] Dennis TA, O'Toole L. Mental Health on the Go: Effects of a Gamified Attention Bias Modification Mobile Application in Trait Anxious Adults. Clin Psychol Sci. 2014 Sep 1;2(5):576-590. doi: 10.1177/2167702614522228. PMID 26029490
- [Result] Escoffery C, McGee R, Bidwell J, Sims C, Thropp EK, Frazier C, Mynatt ED. A review of mobile apps for epilepsy self-management. Epilepsy Behav. 2018 Apr;81:62-69. doi: 10.1016/j.yebeh.2017.12.010. Epub 2018 Mar 20. PMID 29494935
- [Result] Sayik D, Acikgoz A, Yimenicioglu S. A randomized controlled study: Evaluating the efficacy of a mobile application developed for mothers who have children with epilepsy in Turkiye. J Pediatr Nurs. 2023 May-Jun;70:103-110. doi: 10.1016/j.pedn.2023.02.010. Epub 2023 Mar 2. PMID 36870141
- [Result] Wohlrab GC, Rinnert S, Bettendorf U, Fischbach H, Heinen G, Klein P, Kluger G, Jacob K, Rahn D, Winter R, Pfafflin M; Famoses Project Group. famoses: a modular educational program for children with epilepsy and their parents. Epilepsy Behav. 2007 Feb;10(1):44-8. doi: 10.1016/j.yebeh.2006.10.005. Epub 2006 Nov 27. PMID 17126082
- [Result] Turan Gurhopur FD, Isler Dalgic A. The effect of a modular education program for children with epilepsy and their parents on disease management. Epilepsy Behav. 2018 Jan;78:210-218. doi: 10.1016/j.yebeh.2017.07.048. Epub 2017 Dec 6. PMID 29203274